CLINICAL TRIAL: NCT04721522
Title: The Impact of Endometrial Compaction on Assisted Reproductive Technology Outcome
Status: Recruiting | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Rana Nabil Mohamed Attia, Assistant lecturer of obstetrics and gynaecology, Zagazig University
Other Study IDs: 6549
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Embryo Implantation; ART
Keywords: Endometrial Compaction; endometrial receptivity; ART
MeSH Terms: interventions — Blood Specimen Collection; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 356 case will be enrolled: Pituitary suppression will be achieved by long or antagonist protocol. For long protocol, GnRH agonist will be administered for 10-14 days starting from mid-luteal phase of preceding cycle. After confirmation of down regulation, gonadotropins will be given from second or third day of cycle in a daily dose of (150-300 IU). Gonadotropins therapy will be tailored according to age, BMI, antral follicle count, antimullerian hormone and previous response. In antagonist protocol, gonadotropins will be given from second or third day of cycle in a daily dose of (150-300 IU). GnRH antagonist will be adjusted according to patient response. On the 5th -6th day of stimulation, sonography will be performed and repeated every 1-3 days with regular estradiol assessment. When at least 3 follicles reach ≥ 17 mm in mean diameter, trigger will be given. Oocytes pick up will be performed 34-36 hour after triggering.
  Interventions: Diagnostic Test: blood sampling & ultrasound

INTERVENTIONS:
Diagnostic Test: blood sampling & ultrasound — Blood sampling:
  Serum P4 & estradiol will be performed on the day of triggering and on the day of embryo transfer. Progesterone/ Estradiol (P4/E2) ratio will be calculated Ultrasound: On triggering day, at time of ovum pick up and on ET day, we will measure
  1. Endometrial thickness
  2. Endometrial pattern
  3. Endometrial compaction: the difference in measurement of endometrial thickness between the day of embryo transfer and the day of triggering.
  4. Junctional zone thickness
  5. Uterine contraction (peristalsis).
  6. Blood flow of uterine vessels: PI of the uterine arteries will be calculated also Endometrial - sub endometrial blood flow

SUMMARY:
Absence of endometrial compaction on the day of ET has adverse effects on success of ART outcome.

DETAILED DESCRIPTION:
Implantation is a complex process which requires coordination and interaction between a blastocyst and the endometrium. Impaired embryo quality or impaired endometrial receptivity may negatively affect this interaction that in turn results in implantation failure (Diedrich et al., 2007). . Successful implantation entails a process of strict synchronization of endometrial and blastocyst development. (Maged et al., 2018).

Despite advancements made since the introduction of assisted reproductive technology (ART), fewer than 40% of ART treatment cycles result in a live birth. Endometrial receptivity remains a crucial rate-limiting step affecting the success of ART treatment. Embryos are thought to be responsible for one-third of implantation failures, whereas the remaining two-thirds result from sub-optimal endometrial receptivity or abnormal embryo-endometrium dialogue.(Craciunas et al., 2019).

There are 3 main methods used to assess endometrial receptivity: endometrial biopsy, hormone profile, and ultrasound imaging.(Lawrenz and Fatemi, 2017). Ultrasound has been established as an appreciated, simple, and non-invasive technique in evaluation of endometrial preparation before embryo transfer in IVF cycles. Several sonographic parameters have been assessed that include endometrial thickness (Ent), endometrial pattern (EnP) and sub-endometrial blood flow.(Kader et al., 2016).

Endometrial thickness (EMT) is the most used prognostic factor for endometrial receptivity during ART (Kasius et al., 2014). Both clinical pregnancy and live birth rates decreased significantly for each millimeter below 8 mm in fresh IVF-ET cycles and below 7 mm frozen ET cycles (Liu et al 2018). Regarding endometrial patterns (Yuan et al., 2016) and vascularization (Ng et al., 2007) data are still contradictory. Increased frequency of contractility prior to embryo transfer was inversely related to clinical pregnancy in fresh and frozen embryo transfer cycles. (Zhu et al., 2014).

Currently, there is an emphasis on a new endometrial parameter called endometrial compaction, which is the decrease in endometrial thickness on the day of ET. In a Study of 274 frozen embryo transfer cycles, patients whose endometrium compacted had a significantly higher ongoing pregnancy rate than patients whose endometrium became thicker or did not change.(Haas et al., 2019).

On the other hand, a large-scale cohort study revealed that an increased endometrium thickness after progesterone administration in FET was associated with better pregnancy outcome.(Bu et al., 2019). The role of endometrial compaction in fresh ART cycles is not yet studied. So, it's better to test its effect on fresh cycles ART outcome.

ELIGIBILITY:
Inclusion Criteria:

* All women should have the following:

Aged from 18 - 37 years old. Undergoing fresh ICSI cycles. A normal uterus with no anomalies or pathologies. At least one good-quality embryo/blastocyst available for transfer (3 BB and more according to Gardner and Schoolcraft grading system).

Easy mockup embryo transfer (i.e. the catheter is smoothly inserted without touching the fundus, no cervix tenaculum is used and the catheter is clean of blood).

Exclusion Criteria:

- Younger than 18 or older than 37 years old. Congenital uterine abnormality or pathology. Presence of a hydrosalpinx. Chronic diseases which are not suitable for pregnancy. ICSI cycles with fresh or frozen TESE samples.

Ages: 18 Years to 37 Years | Sex: Female
Age Groups: Adult
Study Population: It will be carried out in the department of Obstetrics and Gynecology, Zagazig University and in a private center.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
whether the occurrence of endometrial compaction on the day of embryo transfer has a role in optimizing ongoing pregnancy rate in ART cycles | 2 weeks
  Percent of endometrial compaction will be calculated as the difference in measurement of endometrial thickness between the day of embryo transfer and the day of triggering.

CONTACTS AND LOCATIONS:
Overall Officials: rana nabil, Msc, Principal Investigator — zagazig university hospital
Locations (1):
- Zagazig university, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Diedrich K, Fauser BC, Devroey P, Griesinger G; Evian Annual Reproduction (EVAR) Workshop Group. The role of the endometrium and embryo in human implantation. Hum Reprod Update. 2007 Jul-Aug;13(4):365-77. doi: 10.1093/humupd/dmm011. Epub 2007 Jun 4. PMID 17548368
- [Background] Maged AM, Rashwan H, AbdelAziz S, Ramadan W, Mostafa WAI, Metwally AA, Katta M. Randomized controlled trial of the effect of endometrial injury on implantation and clinical pregnancy rates during the first ICSI cycle. Int J Gynaecol Obstet. 2018 Feb;140(2):211-216. doi: 10.1002/ijgo.12355. Epub 2017 Nov 18. PMID 29048754
- [Background] Craciunas L, Gallos I, Chu J, Bourne T, Quenby S, Brosens JJ, Coomarasamy A. Conventional and modern markers of endometrial receptivity: a systematic review and meta-analysis. Hum Reprod Update. 2019 Mar 1;25(2):202-223. doi: 10.1093/humupd/dmy044. PMID 30624659
- [Background] Lawrenz B, Fatemi HM. Effect of progesterone elevation in follicular phase of IVF-cycles on the endometrial receptivity. Reprod Biomed Online. 2017 Apr;34(4):422-428. doi: 10.1016/j.rbmo.2017.01.011. Epub 2017 Jan 24. PMID 28162937
- [Background] Kader MA, Abdelmeged A, Mahran A, Samra MFA, Bahaa H (2016) The usefulness of endometrial thickness, morphology, and vasculature by 2D Doppler ultrasound in prediction of pregnancy in IVF/ICSI cycles. Egypt J Radiol Ncl Med 47(1):341-346.
- [Background] Kasius A, Smit JG, Torrance HL, Eijkemans MJ, Mol BW, Opmeer BC, Broekmans FJ. Endometrial thickness and pregnancy rates after IVF: a systematic review and meta-analysis. Hum Reprod Update. 2014 Jul-Aug;20(4):530-41. doi: 10.1093/humupd/dmu011. Epub 2014 Mar 23. PMID 24664156
- [Background] Liu KE, Hartman M, Hartman A, Luo ZC, Mahutte N. The impact of a thin endometrial lining on fresh and frozen-thaw IVF outcomes: an analysis of over 40 000 embryo transfers. Hum Reprod. 2018 Oct 1;33(10):1883-1888. doi: 10.1093/humrep/dey281. PMID 30239738
- [Background] Yuan X, Saravelos SH, Wang Q, Xu Y, Li TC, Zhou C. Endometrial thickness as a predictor of pregnancy outcomes in 10787 fresh IVF-ICSI cycles. Reprod Biomed Online. 2016 Aug;33(2):197-205. doi: 10.1016/j.rbmo.2016.05.002. Epub 2016 May 13. PMID 27238372
- [Background] Ng EH, Chan CC, Tang OS, Yeung WS, Ho PC. Endometrial and subendometrial vascularity is higher in pregnant patients with livebirth following ART than in those who suffer a miscarriage. Hum Reprod. 2007 Apr;22(4):1134-41. doi: 10.1093/humrep/del458. Epub 2006 Dec 5. PMID 17148577
- [Background] Zhu L, Che HS, Xiao L, Li YP. Uterine peristalsis before embryo transfer affects the chance of clinical pregnancy in fresh and frozen-thawed embryo transfer cycles. Hum Reprod. 2014 Jun;29(6):1238-43. doi: 10.1093/humrep/deu058. Epub 2014 Mar 23. PMID 24664129
- [Background] Haas J, Smith R, Zilberberg E, Nayot D, Meriano J, Barzilay E, Casper RF. Endometrial compaction (decreased thickness) in response to progesterone results in optimal pregnancy outcome in frozen-thawed embryo transfers. Fertil Steril. 2019 Sep;112(3):503-509.e1. doi: 10.1016/j.fertnstert.2019.05.001. Epub 2019 Jun 24. PMID 31248618
- [Background] Bu Z, Yang X, Song L, Kang B, Sun Y. The impact of endometrial thickness change after progesterone administration on pregnancy outcome in patients transferred with single frozen-thawed blastocyst. Reprod Biol Endocrinol. 2019 Nov 25;17(1):99. doi: 10.1186/s12958-019-0545-0. PMID 31767010